CLINICAL TRIAL: NCT02342301
Title: Cardiometabolic Response to Sit-stand Workstations.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Prince Edward Island (Other)
Responsible Party: Principal Investigator, Travis Saunders, Assistant Professor, University of Prince Edward Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6005871
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standing Desk (Experimental): Will use standing desk for 3 months
  Interventions: Behavioral: Standing Desk
- Traditional Desk (Active Comparator): Will use traditional desk for 3 months
  Interventions: Behavioral: Traditional Desk

INTERVENTIONS:
Behavioral: Standing Desk — Participants will be provided with a standing desk for 3 months
  Arms: Standing Desk
Behavioral: Traditional Desk — Participants will use a traditional seated desk for 3 months
  Arms: Traditional Desk

SUMMARY:
We aim to determine if changing a person's workstation from a traditional seated desk to a height adjustable "standing desk" for a period of approximately 3 months is associated with alterations in traditional measures of cardiometabolic risk.

DETAILED DESCRIPTION:
The present study will include 24 male and female participants 18 years of age and older who work in an office-based setting. To be included participants must be abdominally obese, defined as a waist circumference ≥ 88 cm for women, and 102 cm for men. All potential participants will be asked to come to the Human Performance Laboratory at University of Prince Edward Island and will be given an opportunity to ask questions about the study, and to read and sign the informed consent form. Once this has taken place, participants will have their waist circumference measured in order to determine whether they meet the above criteria. If not, the individual will be thanked for their time and told that they are not eligible to participate in the current study.

Lab Day 1 (baseline)

Once screening is complete, participants will have glycosylated hemoglobin checked via a simple finger prick and point-of-care analysis of a single drop of blood. (Funding dependent, a second drop of blood may be used to analyze the participant's blood lipid profile- as would be done at a typical doctor's office visit). Next we will measure the participants' resting metabolic rate, by having them lay on a hospital bed while we analyze the oxygen and carbon dioxide concentrations of the air they exhale. This will inform us as to the participant's baseline caloric needs. Blood pressure, height, weight, waist circumference and body composition will be determined following resting metabolic rate, prior to the determination of aerobic fitness using a sub-maximal exercise protocol (see below).

Augmentation Index:

Arterial stiffness will be determined using a Sphygmocor pulse wave applanation tonomoter (Atcor Medical). This device measures arterial pulse waves non-invasively through the skin at the wrist. We will use this same device to analyze the shape of the pulse wave, which will give us information about reflected pulse waves (and thus the stiffness of the arterial tree). The measure of arterial stiffness is non-invasive and pain-free and is taken using a pen-like tool pressed against the participant's skin to detect his or her pulse.

Prior to departing the lab, participants will be instructed on the use of an accelerometer-based activity monitor (20 min), which they will wear for 1 week prior to the desk intervention. During the activity monitor collection week, participants will also be instructed to wear a heart rate belt (non-invasive chest strap) for one day during working hours only (at least 4 hours of data collection) which will be analyzed after the strap is returned to the lab. Participants will then answer an online questionnaire about his/her current physical activity and sedentary behaviors. https://docs.google.com/forms/d/1fjz5ua47KzcdnhCAN7wCDGNbvy-tKSGgZKGGhIKSqQg/viewform?usp=mail_form_link . A similar questionnaire will be used for post- intervention follow-up with the tenses changed and questions about "anticipated" desk use altered to report on "actual" use (participants in the control group will be asked to answer "not applicable" for any questions related to standing desk use on the follow-up questionnaire).

Total participation Time (1.5 hr)

Once the baseline testing session is complete, participants will be randomly allocated to intervention or control groups (12 participants per group). Participants in the intervention group will be asked to complete the below intervention, while those in the control group will be asked to maintain their current lifestyle and office workstation throughout the study.

Intervention- the participant will be given a stand-up desk and asked to use it in place of their normal desk at work. Participants will again be given the activity and HR monitors to wear during the first and last 2 weeks of desk use.

Lab day 2 (post) - all measures from lab day 1 will be repeated as described above.

Aerobic Fitness- Aerobic fitness will be determined using a treadmill-based graded exercise test with analysis of expired gases. The test will consist of 2-3 increasingly more challenging stages of walking/running (through the addition of speed or incline) at a submaximal intensity. The heart rate and oxygen consumption data collected will be used to extrapolate the data to estimate maximal values. All aerobic fitness tests will be administered under the supervision of a Canadian Society for Exercise Physiology Certified Exercise Physiologist. Prior to any exercise all participants will be required to complete a Physical Activity Readiness Questionnaire (PAR-Q+) safe exercise participation screening form for known or suspected chronic disease risk factors (this tool is used for screening purposes only).

Resting metabolic rate will be determined using the same electrochemical analyzers (on the same metabolic cart) as the exercise measures, except a different flowmeter and gas collection system will be used (namely, we will use a canopy rather than a face mask). This will allow the participant to relax and rest normally without the need of having their nose and mouth covered by a rubber mask, as their entire head and shoulders will be contained within a canopy to collect gases. This system is identical to those used in-hospital.

ELIGIBILITY:
Inclusion Criteria:

* male and female participants
* 18 years of age and older
* work in an office-based setting.
* abdominally obese, defined as a waist circumference ≥ 88 cm for women, and 102 cm for men.

Exclusion Criteria:

* glucose lowering medication
* inability to stand or walk

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Glycoslyated Hemoglobin (HbA1C) | 3 months
  HbA1c will be measured at baseline and 3 months in both conditions in all participants using a bench-top analyzer.

SECONDARY OUTCOMES:
Sedentary Time | 3 months
  Sedentary time will be measured at baseline and 3 months using an activPAL inclinometer.
Aerobic Fitness (VO2max) | 3 months
  Aerobic Fitness will be measured at baseline and 3 months using a sub-maximal fitness test.
Augmentation Index | 3 months
  Augmentation Index will be measured at baseline and 3 months using a Sphygmocor pulse wave applanation tonomoter.
Waist Circumference | 3 months
  Waist circumference will be measured at baseline and 3 months at the level of the iliac crest.
Physical Activity | 3 months
  Physical activity will be measured at baseline and 3 months using an activPAL inclinometer.
Triglycerides | 3 months
  Plasma triglycerides will be measured at baseline and at 3 months using a bench top analyzer.
Fasting Glucose | 3 months
  Fasting glucose will be measured at baseline and at 3 months using a bench top analyzer.
LDL Cholesterol | 3 months
  LDL Cholesterol will be measured at baseline and at 3 months using a bench top analyzer.
HDL Cholesterol | 3 months
  HDL Cholesterol will be measured at baseline and at 3 months using a bench top analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Burr, PhD, Principal Investigator — University of Prince Edward Island
Locations (1):
- Human Performance and Health Research Lab, University of Prince Edward Island, Charlottetown, Prince Edward Island, Canada

IPD SHARING:
Plan to Share IPD: No